CLINICAL TRIAL: NCT01757535
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Compare Efficacy and Safety of Oral Azacitidine Plus Best Supportive Care Versus Best Supportive Care as Maintenance Therapy in Subjects With Acute Myeloid Leukemia in Complete Remission
Brief Title: Efficacy of Oral Azacitidine Plus Best Supportive Care as Maintenance Therapy in Subjects With Acute Myeloid Leukemia (AML) in Complete Remission
Acronym: QUAZAR AML-001
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-486-AML-001; 2012-003457-28 (EudraCT Number)
Record Dates: First submitted 2012-11-21; First posted 2012-12-31 (Estimated); Results first posted 2020-11-06 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Maintenance therapy; AML; Acute Myeloid Leukemia; Oral Azacitidine; Best supportive care; Complete remission
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Pathologic Complete Response | interventions — Azacitidine; cc-486

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Azacitidine (Experimental): 300 mg oral azacitidine on days 1 to 14 of each 28-day treatment cycle.
  Interventions: Drug: Oral Azacitidine
- Placebo (Placebo Comparator): Identically matching placebo tablets on days 1 to 14 of each 28-day treatment cycle.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral Azacitidine — 300 mg oral azacitidine on days 1 to 14 of each 28-day treatment cycle.
  Other Names: CC-486; Onureg®
  Arms: Oral Azacitidine
Drug: Placebo — Identically matching placebo tablets on days 1 to 14 of each 28-day treatment cycle.
  Arms: Placebo

SUMMARY:
This study enrolled 472 participants, aged 55 or older, with a diagnosis of de novo acute myeloid leukemia (AML) or AML secondary to prior myelodysplastic disease or chronic myelomonocytic leukemia (CMML), and who have achieved first complete remission (CR)/ complete remission with incomplete blood count recovery (CRi) following induction with or without consolidation chemotherapy.

The study is amended to include an extension phase (EP). The EP allows participants who are currently receiving oral azacitidine and who are demonstrating clinical benefit as assessed by the investigator, to continue receiving oral azacitidine after unblinding by sponsor until the participant meets the criteria for study discontinuation or until oral azacitidine becomes commercially available and reimbursed. In addition, all participants in the placebo arm and participants who had been discontinued from the treatment phase (irrespective of randomization arm) and continuing in the follow-up phase will be followed for survival in the EP.

DETAILED DESCRIPTION:
This is an international, multicenter, placebo-controlled, Phase 3 study with a double-blind, randomized, parallel-group design in subjects with de novo AML or AML secondary to prior diagnosis of myelodysplastic syndromes (MDS) or chronic myelomonocytic leukemia (CMML) aged ≥ 55 years, who are in first CR/CRi following induction therapy with or without consolidation chemotherapy. The study consists of 3 phases; the pre-randomization phase (screening phase), the treatment phase, and the follow-up phase.

The study is amended to include an extension phase (EP). The EP allows participants who are currently receiving oral azacitidine and who are demonstrating clinical benefit as assessed by the Investigator, to continue receiving oral azacitidine after unblinding by sponsor until they meet the criteria for study discontinuation or until oral azacitidine becomes commercially available and reimbursed. In addition, all participants in the placebo arm and participants who had been discontinued from the treatment phase (irrespective of randomization arm) and continuing in the follow-up phase will be followed for survival in the EP.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female participants ≥ 55 years of age
2. Newly diagnosed, histologically confirmed de novo acute myeloid leukemia (AML) or AML secondary to prior myelodysplastic disease or CMML (Chronic myelomonocytic leukemia)
3. First complete remission (CR)/ complete remission with incomplete blood count recovery (CRi) with induction therapy with intensive chemotherapy with or without consolidation therapy within 4 months (+/- 7 days of achieving CR or CRi)
4. Eastern Cooperative Oncology Group (ECOG) performance status - 0, 1, 2, 3

Key Inclusion Criteria in the Extended Phase of the study:

At the Investigator's discretion and with approval of the sponsor, participants meeting all of the following eligibility criteria are eligible to enter the extension phase:

1. All participants randomized into the oral azacitidine or placebo arm and are continuing in either the treatment phase or follow-up phase of the CC-486-AML-001 study;

   * Participants randomized to oral azacitidine treatment arm and continuing in the treatment phase demonstrating clinical benefit as assessed by the investigator are eligible to receive oral azacitidine in the extension phase (EP);
   * Participants randomized into placebo arm of the study will not receive oral azacitidine in the EP, but will be followed for survival in the EP;
   * Participants currently in the follow-up phase will continue to be followed for survival in the EP;
2. Participants who have signed the informed consent for the EP of the study;
3. Participants who do not meet any of the criteria for study discontinuation

Key Exclusion Criteria:

1. AML with inversion (inv)(16), translocation = t(8;21), t(16;16), t(15;17), or t(9;22) or molecular evidence of such translocations
2. Prior bone marrow or stem cell transplantation
3. Have achieved CR/CRi following therapy with hypomethylating agents
4. Diagnosis of malignant disease within the previous 12 months
5. Proven central nervous system (CNS) leukemia

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2013-04-24 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2024-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (223):
- United States (60):
  - Arizona Oncology Associates, P.C., Phoenix, Arizona
  - Providence St Joseph Medical Center Cancer Center, Burbank, California
  - City Of Hope, Duarte, California
  - University of California San Francisco Fresno Campus, Fresno, California
  - University of Southern California Norris Cancer Center, Los Angeles, California
  - Local Institution - 006, Los Angeles, California
  - Local Institution - 050, Orange, California
  - Sharp Memorial Hospital, San Diego, California
  - Stanford Cancer Center, Stanford, California
  - Innovative Clinical Research Institute, Whittier, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Local Institution - 010, Southington, Connecticut
  - George Washington University Cancer Center, Washington D.C., District of Columbia
  - Local Institution - 046, Gainesville, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Local Institution - 044, Orlando, Florida
  - Northwestern University Medical Center, Chicago, Illinois
  - Loyola University Chicago, Maywood, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland, P.C. - Niles, IL, Niles, Illinois
  - Local Institution - 013, Indianapolis, Indiana
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - Local Institution - 003, Westwood, Kansas
  - Local Institution - 049, Louisville, Kentucky
  - Local Institution - 058, Louisville, Kentucky
  - Local Institution - 047, New Orleans, Louisiana
  - Ochsner Medical Center - Jefferson Highway, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Local Institution - 015, Worcester, Massachusetts
  - Local Institution - 037, Rochester, Minnesota
  - Local Institution - 023, Kansas City, Missouri
  - Washington University School Of Medicine, St Louis, Missouri
  - Local Institution - 057, Omaha, Nebraska
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - Local Institution - 009, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Local Institution - 002, New York, New York
  - Local Institution - 004, Rochester, New York
  - Local Institution - 014, Valhalla, New York
  - Duke University Medical Center, Durham, North Carolina
  - Local Institution - 025, Winston-Salem, North Carolina
  - Local Institution - 016, Cleveland, Ohio
  - University of Oklahoma Peggy and Charles Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Kaiser Permanente Northwest Oncology Hematology, Portland, Oregon
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - UPMC Cancer Pavillion, Pittsburgh, Pennsylvania
  - Greenville Hospital System, Greenville, South Carolina
  - Local Institution - 011, Nashville, Tennessee
  - Local Institution - 007, Nashville, Tennessee
  - Local Institution - 041, Dallas, Texas
  - Local Institution - 034, Fort Sam Houston, Texas
  - Local Institution - 001, Houston, Texas
  - Cancer Care Centers of South Texas - Loop, San Antonio, Texas
  - Local Institution - 039, San Antonio, Texas
  - Local Institution - 035, Richmond, Virginia
  - Swedish Cancer Inst, Seattle, Washington
  - Yakima Valley Memorial Hospital/ North Star Lodge, Yakima, Washington
  - Froedtert Hospital BMT Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (13):
  - Local Institution - 510, Wollongong, New South Wales
  - Local Institution - 509, South Brisbane, Queensland
  - Local Institution - 508, Adelaide, South Australia
  - Local Institution - 511, Bedford Park, South Australia
  - Local Institution - 504, Woodville South, South Australia
  - Local Institution - 503, Heidelberg
  - Local Institution - 502, Hobart
  - Local Institution - 507, Liverpool
  - Local Institution - 500, Melbourne
  - Local Institution - 505, Perth
  - Local Institution - 512, Perth
  - Local Institution - 506, St Leonards
  - Local Institution - 501, Woolloongabba
- Austria (5):
  - Local Institution - 271, Graz
  - Local Institution - 270, Salzburg
  - Local Institution - 274, Vienna
  - Local Institution - 272, Vienna
  - Local Institution - 273, Vienna
- Belgium (3):
  - Local Institution - 300, Bruges
  - Local Institution - 301, Charleroi
  - Local Institution - 302, Mons
- Brazil (5):
  - Local Institution - 233, Curitiba, Paraná
  - Local Institution - 231, Porto Alegre, Rio Grande do Sul
  - Local Institution - 232, Rio de Janeiro
  - Local Institution - 234, São Paulo
  - Local Institution - 230, São Paulo
- Canada (8):
  - Local Institution - 605, Edmonton, Alberta
  - Local Institution - 600, Winnipeg, Manitoba
  - Local Institution - 601, Saint John, New Brunswick
  - Local Institution - 603, St. John's, Newfoundland and Labrador
  - Local Institution - 604, Halifax, Nova Scotia
  - Local Institution - 607, Toronto, Ontario
  - Local Institution - 608, Montreal, Quebec
  - Local Institution - 602, Montreal, Quebec
- Czechia (3):
  - Local Institution - 320, Brno, South Moravian
  - Local Institution - 321, Prague
  - Local Institution - 322, Prague
- Finland (3):
  - Local Institution - 361, Helsinki
  - Local Institution - 362, Tampere
  - Local Institution - 360, Turku
- France (17):
  - Local Institution - 456, Amiens
  - Local Institution - 465, Argenteuil
  - Local Institution - 457, Bobigny
  - Local Institution - 462, Boulognes Sur Mer
  - Local Institution - 460, Clamart
  - Local Institution - 452, Créteil
  - Local Institution - 458, Le Chesnay
  - Local Institution - 453, Lille
  - Local Institution - 461, Limoges
  - Local Institution - 450, Lyon
  - Local Institution - 463, Paris
  - Local Institution - 454, Paris
  - Local Institution - 800, Paris
  - Local Institution - 464, Pontoise
  - Local Institution - 455, Rouen
  - Local Institution - 459, Saint-Cloud
  - Local Institution - 451, Villejuif
- Germany (17):
  - Local Institution - 400, Dresden, Saxony
  - Local Institution - 413, Berlin
  - Local Institution - 410, Bonn
  - Local Institution - 406, Düsseldorf
  - Local Institution - 415, Erlangen
  - Local Institution - 404, Frankfurt am Main
  - Local Institution - 412, Goch
  - Local Institution - 405, Hanover
  - Local Institution - 408, Heilbronn
  - Local Institution - 414, Jena
  - Local Institution - 403, Keil
  - Local Institution - 402, Mannheim
  - Local Institution - 409, München
  - Local Institution - 411, München
  - Local Institution - 407, Oldenburg
  - Local Institution - 416, Schweiler
  - Local Institution - 401, Ulm
- Ireland (2):
  - Local Institution - 950, Dublin
  - Local Institution - 951, Galway
- Israel (4):
  - Local Institution - 381, Beersheba
  - Local Institution - 380, Haifa
  - Local Institution - 383, Jerusalem
  - Local Institution - 382, Petah Tikva
- Italy (26):
  - Local Institution - 701, Alessandria
  - Local Institution - 721, Bari
  - Local Institution - 720, Bologna
  - Local Institution - 710, Cagliari
  - Local Institution - 702, Cremona
  - Local Institution - 708, Florence
  - Local Institution - 712, Genova
  - Local Institution - 716, Lecce
  - Local Institution - 706, Milan
  - Local Institution - 726, Milan
  - Local Institution - 704, Monza
  - Local Institution - 717, Naples
  - Local Institution - 725, Naples
  - Local Institution - 705, Orbassano (TO)
  - Local Institution - 703, Palermo
  - Local Institution - 719, Palermo
  - Local Institution - 724, Pesaro
  - Local Institution - 700, Reggio Calabria
  - Local Institution - 709, Roma
  - Local Institution - 714, Roma
  - Local Institution - 723, Roma
  - Local Institution - 722, Rome
  - Local Institution - 715, Torino
  - Local Institution - 718, Torino
  - Local Institution - 711, Udine
  - Local Institution - 707, Varese
- Local Institution - 750, Klaipėda, Lithuania
- Mexico (3):
  - Local Institution - 252, Huixquilucan de Degollado
  - Local Institution - 251, México
  - Local Institution - 250, Monterrey
- Poland (5):
  - Local Institution - 824, Bydgoszcz
  - Local Institution - 820, Gdansk
  - Local Institution - 822, Lodz
  - Local Institution - 821, Warsaw
  - Local Institution - 823, Wroclaw
- Portugal (5):
  - Local Institution - 841, Coimbra
  - Local Institution - 840, Lisbon
  - Local Institution - 843, Lisbon
  - Local Institution - 842, Porto
  - Local Institution - 844, Porto
- Russia (4):
  - Local Institution - 971, Moscow
  - Local Institution - 970, Nizhny Novgorod
  - Local Institution - 972, Saint Petersburg
  - Local Institution - 973, Saint Petersburg
- South Korea (6):
  - Local Institution - 535, Busan
  - Local Institution - 533, Daegu
  - Local Institution - 536, Seoul
  - Local Institution - 530, Seoul
  - Local Institution - 531, Seoul
  - Local Institution - 532, Seoul
- Spain (14):
  - Local Institution - 872, Palma de Mallorca, Balearic Islands
  - Local Institution - 867, A Coruña
  - Local Institution - 869, Badalona (Barcelona)
  - Local Institution - 871, Barcelona
  - Local Institution - 870, Barcelona
  - Local Institution - 873, Cáceres
  - Local Institution - 863, Córdoba
  - Local Institution - 868, Madrid
  - Local Institution - 866, Madrid
  - Local Institution - 865, Madrid
  - Local Institution - 864, Oviedo
  - Local Institution - 861, Salamanca
  - Local Institution - 862, Seville
  - Local Institution - 860, Valencia
- Taiwan (5):
  - Local Institution - 599, Beitou District, Taipei City
  - Local Institution - 595, Niaosong District Kaohsiung City
  - Local Institution - 596, Taichung, Northern Dist.
  - Local Institution - 597, Tainan, Taiana
  - Local Institution - 598, Taipei, Zhongzheng Dist.
- Turkey (Türkiye) (4):
  - Local Institution - 653, Ankara
  - Local Institution - 650, Ankara
  - Local Institution - 651, Istanbul
  - Local Institution - 652, Samsun
- United Kingdom (10):
  - Local Institution - 904, Nottingham, Nottinghamshire
  - Local Institution - 907, Boston
  - Local Institution - 903, Brighton East Sussex
  - Local Institution - 902, Canterbury Kent
  - Local Institution - 905, London
  - Local Institution - 901, London
  - Local Institution - 908, London
  - Local Institution - 909, Maidstone
  - Local Institution - 900, Manchester
  - Local Institution - 906, Romford, Essex

REFERENCES:
- [Background] Roboz GJ, Montesinos P, Selleslag D, Wei A, Jang JH, Falantes J, Voso MT, Sayar H, Porkka K, Marlton P, Almeida A, Mohan S, Ravandi F, Garcia-Manero G, Skikne B, Kantarjian H. Design of the randomized, Phase III, QUAZAR AML Maintenance trial of CC-486 (oral azacitidine) maintenance therapy in acute myeloid leukemia. Future Oncol. 2016 Feb;12(3):293-302. doi: 10.2217/fon.15.326. Epub 2016 Jan 19. PMID 26785287
- [Derived] Ravandi F, Dohner H, Wei AH, Montesinos P, Pfeilstocker M, Papayannidis C, Lai Y, Wang K, See WL, de Menezes DL, Petrlik E, Prebet T, Roboz GJ. Survival outcomes in patients with acute myeloid leukaemia who received subsequent therapy for relapse in QUAZAR AML-001. Br J Haematol. 2024 Mar;204(3):877-886. doi: 10.1111/bjh.19202. Epub 2023 Nov 12. PMID 37952982
- [Derived] Wei AH, Roboz GJ, Dombret H, Dohner H, Schuh AC, Montesinos P, Selleslag D, Bondarenko SN, Prebet T, Lai Y, Skikne B, Beach CL, Ravandi F. Survival outcomes with oral azacitidine maintenance in patients with acute myeloid leukemia in remission by receipt of initial chemotherapy: subgroup analyses from the phase III QUAZAR AML-001 trial. Haematologica. 2023 Oct 1;108(10):2820-2825. doi: 10.3324/haematol.2022.282296. No abstract available. PMID 36951156
- [Derived] Dohner H, Wei AH, Roboz GJ, Montesinos P, Thol FR, Ravandi F, Dombret H, Porkka K, Sandhu I, Skikne B, See WL, Ugidos M, Risueno A, Chan ET, Thakurta A, Beach CL, Lopes de Menezes D. Prognostic impact of NPM1 and FLT3 mutations in patients with AML in first remission treated with oral azacitidine. Blood. 2022 Oct 13;140(15):1674-1685. doi: 10.1182/blood.2022016293. PMID 35960871
- [Derived] Zhu J, Wu Q, Wang J, Niu T. Cost-effectiveness analysis of azacitidine maintenance therapy in patients with acute myeloid leukemia. Expert Rev Hematol. 2022 Apr;15(4):375-382. doi: 10.1080/17474086.2022.2061456. Epub 2022 May 11. PMID 35437111
- [Derived] Roboz GJ, Ravandi F, Wei AH, Dombret H, Thol F, Voso MT, Schuh AC, Porkka K, La Torre I, Skikne B, Zhong J, Beach CL, Risueno A, Menezes DL, Ossenkoppele G, Dohner H. Oral azacitidine prolongs survival of patients with AML in remission independently of measurable residual disease status. Blood. 2022 Apr 7;139(14):2145-2155. doi: 10.1182/blood.2021013404. PMID 34995344
- [Derived] Ravandi F, Roboz GJ, Wei AH, Dohner H, Pocock C, Selleslag D, Montesinos P, Sayar H, Musso M, Figuera-Alvarez A, Safah H, Tse W, Sohn SK, Hiwase D, Chevassut T, Pierdomenico F, La Torre I, Skikne B, Bailey R, Zhong J, Beach CL, Dombret H. Management of adverse events in patients with acute myeloid leukemia in remission receiving oral azacitidine: experience from the phase 3 randomized QUAZAR AML-001 trial. J Hematol Oncol. 2021 Aug 28;14(1):133. doi: 10.1186/s13045-021-01142-x. PMID 34454540
- [Derived] Wei AH, Dohner H, Pocock C, Montesinos P, Afanasyev B, Dombret H, Ravandi F, Sayar H, Jang JH, Porkka K, Selleslag D, Sandhu I, Turgut M, Giai V, Ofran Y, Kizil Cakar M, Botelho de Sousa A, Rybka J, Frairia C, Borin L, Beltrami G, Cermak J, Ossenkoppele GJ, La Torre I, Skikne B, Kumar K, Dong Q, Beach CL, Roboz GJ; QUAZAR AML-001 Trial Investigators. Oral Azacitidine Maintenance Therapy for Acute Myeloid Leukemia in First Remission. N Engl J Med. 2020 Dec 24;383(26):2526-2537. doi: 10.1056/NEJMoa2004444. PMID 33369355
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 472 Participants Randomized, 469 participants treated
Groups:
- Oral Azacitidine Plus Best Supportive Care: Participants received 300 mg azacitidine tablets once a day (QD) for the first 14 days of each 28-day treatment cycle until discontinuation, which includes the following reasons: disease relapse, withdrawal of consent, adverse events, participant became eligible for allogeneic bone marrow or stem cell transplantation during the treatment period, death, lost to follow-up, or protocol violation or until the end of the study.
- Placebo Plus Best Supportive Care: Participants received identically matching placebo tablets QD for the first 14 days of each 28-day treatment cycle until no longer receiving benefit, withdrawal of consent, disease relapse, adverse events, participant became eligible for allogeneic bone marrow or stem cell transplantation during the treatment period, lost to follow-up, or protocol violation or until the end of the study.
Period: Overall Study
Arm/Group | Oral Azacitidine Plus Best Supportive Care | Placebo Plus Best Supportive Care
Started (Treatment Phase) | 238 | 234
Received Treatment | 236 | 233
Completed | 0 | 0
Not Completed | 238 | 234
Not completed — Disease Relapse | 151 | 181
Not completed — Other Reasons | 28 | 27
Not completed — Adverse Event | 31 | 11
Not completed — Withdrew Consent | 19 | 13
Not completed — Physician Decision | 7 | 0
Not completed — Death | 2 | 2

BASELINE CHARACTERISTICS:
Population: The intent to treat (ITT) population includes participants who were randomized, regardless of whether they received treatment or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Azacitidine Plus Best Supportive Care | Placebo Plus Best Supportive Care | Total
Number analyzed (Participants) | 238 | 234 | 472
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.9 (5.72) | 68.0 (5.62) | 67.9 (5.66)
Age, Customized [Count of Participants; unit: Participants]
  18 to 64 Years | 66 | 68 | 134
  65 to 84 Years | 171 | 166 | 337
  ≥ 85 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 107 | 227
  Male | 118 | 127 | 245
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 14 | 34
  Not Hispanic or Latino | 196 | 202 | 398
  Unknown or Not Reported | 22 | 18 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 216 | 197 | 413
  Black or African-American | 2 | 6 | 8
  Asian | 6 | 20 | 26
  Other | 12 | 11 | 23
  Missing | 2 | 0 | 2
Initial Acute Myeloid Leukemia (AML) Classification [Count of Participants; unit: Participants] — AML is classified using the WHO classification system based upon a combination of morphology, immunophenotype, genetics, and clinical features. There are several broad groups and include: 1. AML with genetic abnormalities; 2. AML with multilineage dysplasia 3. AML related to previous chemotherapy or radiation 4. Unspecified AML - do not fall into the above groups
  Participants
    AML with Recurrent Genetic Abnormalities | 39 | 46 | 85
    AML with Myelodysplasia - Related Changes | 49 | 42 | 91
    Therapy-related Myeloid Neoplasms | 2 | 0 | 2
    AML not Otherwise Specified | 148 | 145 | 293
    Missing | 0 | 1 | 1
Type of Acute Myeloid Leukemia (AML) [Count of Participants; unit: Participants] — Primary AML is a cancer that originates in the blood and bone marrow. AML affects a group of white blood cells called myeloid cells, which normally develop into the various types of mature blood cells, such as red blood cells, white blood cells and platelets. Secondary acute myeloid leukemia (s-AML) refers to a leukemic process: (1) evolving from prior myelodysplasia (MDS), myeloproliferative disorder (MPN), or aplastic anemia (AA) with or without treatment or (2) as a product of previous exposure to a proven leukemogenic chemotherapeutic agent (therapy-related AML [t-AML]).
  Participants
    Primary (de novo) | 213 | 216 | 429
    Secondary | 25 | 18 | 43
Cytogenetic Risk Category at Diagnosis [Count of Participants; unit: Participants] — Cytogenetic Risk - Intermediate -I is of a normal karyotype; Poor Risk - includes complex karyotypes having 3 or more cytogenetic abnormalities.
  Participants
    Intermediate | 203 | 203 | 406
    Poor | 35 | 31 | 66
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status is used to describe a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.). The scale ranges from 0 to 5: 0 = Fully active, no restrictions; 1 = Restricted activity but ambulatory, able to carry out work of a light nature; 2 = Ambulatory and capable of all self-care but unable to carry out work activities; 3 = Capable to only limited self-care, confined to bed or chair more than 50% of waking hours; 4 = Completely disabled, no self-care, confined to bed or chair; 5 = Dead.
  Participants
    Grade 0 | 116 | 111 | 227
    Grade 1 | 101 | 106 | 207
    Grade 2 | 21 | 15 | 36
    Grade 3 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier (K-M) Estimate for Overall Survival (OS)
Description: Overall survival was defined as time from randomization to death from any cause; participants surviving at the end of the follow-up period, or who withdraw consent, or who were lost to follow up were censored at the date last known alive.
Time Frame: Day 1 (randomization) up to data cut off date of 15 July 2019; median follow-up for OS estimated by the reverse K-M method was 41.2 months for all participants.
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Oral Azacitidine Plus Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 238 | 234
Months | 24.7 [18.7 to 30.5] | 14.8 [11.7 to 17.6]
Statistical Analysis 1: Comparison: Oral Azacitidine Plus Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.0009, Log Rank — The p-value is 2-sided from a log-rank test stratified by age, cytogenetic risk category, and received consolidation therapy or not; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.55 to 0.86] — The hazard ratio is from a Cox proportional hazards model stratified by age, cytogenetic risk category, and received consolidation therapy or not; The confidence interval (CI) for the difference was derived using Kosorok's method

2. Secondary Outcome: Kaplan-Meier Estimate of Relapse Free Survival (RFS)
Description: RFS was defined as the time from the date of randomization to the date of documented relapse or death from any cause, whichever occurred first. Participants who were still alive without documented relapse, or who were lost to follow-up or withdrew consent without documented relapse, were censored at the date of their last bone marrow assessment, prior to receiving any other therapy for AML. Documented relapse was defined as the earliest date of the following: • ≥ 5% bone marrow blasts (myeloblasts) from Central Pathology report, or • appearance of > 0% blasts in the peripheral blood with a later bone marrow confirmation (bone marrow blast [myeloblasts] ≥ 5%) within 100 days, or • at least 2 peripheral blasts ≥ 5% within 30 days.
Time Frame: From day 1 (randomization) up to data cut off date of 06 August 2024; approximately 135.5 months
Population: The intent to treat population includes participants who were randomized, regardless of whether they received treatment or not.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Oral Azacitidine Plus Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 238 | 234
Months | 10.2 [7.9 to 12.9] | 4.8 [4.6 to 6.4]
Statistical Analysis 1: Comparison: Oral Azacitidine Plus Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p < 0.0001, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.52 to 0.80] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Kaplan-Meier Estimate of Time to Relapse
Description: Time to relapse was defined as the interval (in months) from the date of randomization to the date of documented relapse. Estimates of relapse rate were based on the cumulative incidence function from a competing risk analysis with death as a competing risk for relapse from complete remission (CR)/ complete remission with incomplete blood count recovery (CRi). Documented relapse was defined as, the earliest date of the following: • ≥ 5% bone marrow blasts (myeloblasts) from Central Pathology report, or • appearance of > 0% blasts in the peripheral blood with a later bone marrow confirmation (bone marrow blast [myeloblasts] ≥ 5%) within 100 days, or • at least 2 peripheral blasts ≥ 5% within 30 days.
Time Frame: From day 1 (randomization) up to data cut off date of 06 August 2024; approximately 135.5 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Oral Azacitidine Plus Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 238 | 234
months | 10.2 [8.3 to 13.4] | 4.9 [4.6 to 6.4]

4. Secondary Outcome: Kaplan-Meier Estimates of Time to Discontinuation From Treatment
Description: Time to discontinuation from treatment was assessed and defined as the interval from the date of randomization to the date of discontinuation from study drug. Participants who were receiving treatment at the time of study closure were censored at the date of last visit. Estimates of relapse rate were based on the cumulative incidence function from a competing risk analysis with death as a competing risk for relapse from CR/ CRi.
Time Frame: From day 1 (randomization) up to data cut off date of 06 August 2024; approximately 135.5 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Oral Azacitidine Plus Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 238 | 234
months | 14.6 [11.3 to 20.1] | 6.9 [5.3 to 7.9]

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs include AEs that started between first dose date and 28 days after the last dose of study drug. A serious adverse event (SAE) is: • Death • Life-threatening event • Inpatient hospitalization or prolongation of existing hospitalization • Persistent or significant disability or incapacity • Congenital anomaly or birth defect • Other important medical event The severity of AEs were assessed by the investigator according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0: Grade 1 (Mild): asymptomatic/mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 (Moderate): minimal, local or noninvasive intervention indicated; limiting age-appropriate activities of daily living. Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care Grade 4: Life-threatening; urgent intervention indicated. Grade 5: Death due to AE.
Time Frame: From day 1 (randomization) up to data cut off date of 06 August 2024; approximately 135.5 months
Population: The safety population included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Azacitidine Plus Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 236 | 233
Participants
  ≥ 1 TEAE | 235 | 233
  ≥ 1 TEAE Related to Study Treatment | 213 | 121
  ≥ 1 Serious TEAE | 110 | 109
  ≥ 1 Treatment Related Serious TEAE | 22 | 5
  ≥ 1 Grade 3/4 TEAE | 207 | 201
  ≥ 1 Treatment Related Grade 3/4 TEAE | 113 | 55
  ≥ 1 TEAE Leading to Death | 15 | 11
  ≥ 1 TEAE Leading to Dose Reduction (Red) | 37 | 6
  ≥ 1 TEAE Leading to Dose Interruption | 107 | 43
  ≥ 1 TEAE Leading to Dose Red and Interruption | 25 | 3
  ≥ 1 TEAE Leading to Study Drug Discontinuation | 155 | 170

6. Secondary Outcome: Mean Change in the Functional Assessment of Chronic Illness Therapy (FACIT-Fatigue Scale V 4.0) Score From Baseline
Description: The functional assessment of chronic illness therapy (FACIT-Fatigue Scale V 4.0) is a subscale of the FACIT-F and has been validated in the oncology setting. The FACIT-Fatigue Scale is a short, 13-item, self-administered tool that measures the level of fatigue in an individual during usually daily activities over the past week. The level of fatigue is measured on a 5-point Likert scale (0 = not at all; 4 = very much. The scores range from 0 to 52, with higher scores indicating less fatigue. If there were missing items, but the participant answered at least 50% of the items, then subscores were prorated.
Time Frame: From day 1 (randomization) up to data cut off date of 06 August 2024; approximately 135.5 months
Population: All treated participants with FACIT-Fatigue measurement by EOT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oral Azacitidine Plus Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 165 | 150
units on a scale | -3.7 (10.92) | -2.5 (9.93)

7. Secondary Outcome: Mean Change in the European Quality of Life-Five Dimensions-Three Levels (EQ-5D-3L) Score From Baseline
Description: The EQ-5D-3L is a self-administered questionnaire consisting of 5 questions, pertaining to specific health dimensions (ie, mobility, self-care, pain, usual activities, and anxiety/depression) and a health status scale. Each question has 3 levels of severity, corresponding to no problems, moderate problems and severe problems. Canadian population sample weights were used to derive health utility scores. A higher utility score represents a better health state. A clinically meaningful improvement or worsening was defined as at least 0.08 points of improvement or 0.10 points of worsening from baseline, respectively, for the EQ-5D-3L Health Utility Index. The instrument is scored using the United Kingdom (UK) index ranges from -0.594 to 1, where 0 equates to death and 1 equates to full health; -0.594 is considered 'worse than death'.
Time Frame: From day 1 (randomization) up to data cut off date of 06 August 2024; approximately 135.5 months
Population: All treated participants with a EQ-5D-3L measurement at the end of treatment
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Oral Azacitidine Plus Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 164 | 150
Units on a scale | -0.0416 (0.15467) | -0.0152 (0.14799)

8. Secondary Outcome: Time to Definitive Clinically Meaningful Deterioration for ≥ 2 Consecutive Visits as Measured Using the EQ-5D HRQoL Scale
Description: Clinically meaningful deterioration was defined at least 0.10 point of deterioration from baseline for at least 2 consecutive visits for the EQ-5D Health Utility Index. The EQ-5D-3L is a self-administered questionnaire consisting of 5 questions, pertaining to specific health dimensions (ie, mobility, self-care, pain, usual activities, and anxiety/depression) and a health status scale. Each question has 3 levels of severity, corresponding to no problems, moderate problems and severe problems. Canadian population sample weights were used to derive health utility scores. A higher utility score represents a better health state. A clinically meaningful improvement or worsening was defined as at least 0.08 points of improvement or 0.10 points of worsening from baseline, respectively, for the EQ-5D-3L Health Utility Index. The EQ-5D-3L is scored using the UK index ranges from -0.594 to 1, where 0 equates to death and 1 equates to full health; -0.594 is considered 'worse than death'.
Time Frame: From day 1 (randomization) up to data cut off date of 15 July 2019; approximately 74 months
Population: The Health Related Quality of Life (HRQoL) evaluable population was defined as the ITT participants with a non-missing EQ-5D-3L score at baseline (C1D1) and at least one post-baseline visit. Results are presented for each post-baseline visit with sample size ≥ 25 in both arms. Death was censored at the date of the last HRQoL assessment visit.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Oral Azacitidine Plus Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 225 | 217
Weeks | NA [135.1 to NA] — Not estimable because the survival curve does not drop to or below 0.5, i.e. the cumulative probability of developing clinically meaningful deterioration does not reach or exceed 50%, during the observation period | NA [122.9 to NA] — Not estimable because the survival curve does not drop to or below 0.5, i.e. the cumulative probability of developing clinically meaningful deterioration does not reach or exceed 50%, during the observation period
Statistical Analysis 1: Comparison: Oral Azacitidine Plus Best Supportive Care vs Placebo Plus Best Supportive Care; Test type: Superiority; p = 0.7522, Regression, Cox — Stratification factors: • Age (at induction therapy): 55 to 64 years and ≥ 65 years • Prior history of MDS: yes/no • Cytogenetic risk (at induction therapy): intermediate-risk/poor-risk • Received consolidation therapy following induction: yes/no; Hazard Ratio (HR) = 0.9345, 95% CI 2-sided [0.6136 to 1.4231]

9. Secondary Outcome: Healthcare Resource Utilization (HRU): Rate of Hospital Events Per Person Year
Description: HRU is defined as any consumption of healthcare resources directly or indirectly related to the treatment of the patient. HRU is a key component to understand treatment costs and budget impact of new treatments from a provider perspective.
Time Frame: From day 1 (randomization) up to data cut off date of 06 August 2024; approximately 135.5 months
Population: Safety population includes all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Hospitalizations per person-years
Arm/Group | Oral Azacitidine Plus Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 236 | 233
Hospitalizations per person-years | 0.36 [0.31 to 0.42] | 0.63 [0.54 to 0.74]

10. Secondary Outcome: Healthcare Resource Utilization (HRU): Number of Days Hospitalized Per Person-Year
Description: as for outcome 9
Time Frame: From day 1 (randomization) up to data cut off date of 06 August 2024; approximately 135.5 months
Population: Safety population includes all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Days per person-years
Arm/Group | Oral Azacitidine Plus Best Supportive Care | Placebo Plus Best Supportive Care
Number analyzed (Participants) | 236 | 233
Days per person-years | 6.00 [5.78 to 6.22] | 13.13 [12.68 to 13.60]

ADVERSE EVENTS:
Time Frame: From day 1 (randomization) up to data cut off date of 06 August 2024; approximately 135.5 months
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Arm/Group | Oral Azacitidine Plus Best Supportive Care | Placebo Plus Best Supportive Care
All-Cause Mortality (participants affected / at risk) | 172/238 | 176/234
Serious Adverse Events (participants affected / at risk) | 110/236 | 109/233
Other Adverse Events (participants affected / at risk) | 235/236 | 224/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Azacitidine Plus Best Supportive Care (N=236) | Placebo Plus Best Supportive Care (N=233)
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 16 | 9
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Aortic valve disease (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0
Iridocyclitis (Eye disorders) | 1 | 0
Keratitis (Eye disorders) | 1 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0
Gastroenteritis eosinophilic (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Neutropenic colitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 2
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 1
General physical health deterioration (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 2
Pyrexia (General disorders) | 6 | 1
Cholecystitis (Hepatobiliary disorders) | 3 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Allergy to vaccine (Immune system disorders) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 4 | 1
Cholecystitis infective (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 1
Device related sepsis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Endophthalmitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Gastroenteritis Escherichia coli (Infections and infestations) | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 3 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 2 | 2
Osteomyelitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 13 | 7
Pneumonia aspiration (Infections and infestations) | 1 | 1
Pneumonia fungal (Infections and infestations) | 1 | 1
Pseudomonas infection (Infections and infestations) | 1 | 0
Rectal abscess (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 5 | 4
Septic shock (Infections and infestations) | 2 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Superinfection bacterial (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Urinary tract infection bacterial (Infections and infestations) | 2 | 0
Urosepsis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Cataract traumatic (Injury, poisoning and procedural complications) | 0 | 1
Chemical peritonitis (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
General physical condition abnormal (Investigations) | 0 | 1
Troponin increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 37 | 58
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Central nervous system leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gliomatosis cerebri (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Central nervous system inflammation (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 2 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Azacitidine Plus Best Supportive Care (N=236) | Placebo Plus Best Supportive Care (N=233)
Anaemia (Blood and lymphatic system disorders) | 51 | 42
Febrile neutropenia (Blood and lymphatic system disorders) | 14 | 10
Leukopenia (Blood and lymphatic system disorders) | 27 | 19
Neutropenia (Blood and lymphatic system disorders) | 104 | 61
Thrombocytopenia (Blood and lymphatic system disorders) | 81 | 62
Abdominal pain (Gastrointestinal disorders) | 32 | 15
Abdominal pain upper (Gastrointestinal disorders) | 23 | 13
Constipation (Gastrointestinal disorders) | 92 | 56
Diarrhoea (Gastrointestinal disorders) | 119 | 50
Dyspepsia (Gastrointestinal disorders) | 12 | 5
Flatulence (Gastrointestinal disorders) | 12 | 4
Haemorrhoids (Gastrointestinal disorders) | 12 | 4
Nausea (Gastrointestinal disorders) | 153 | 54
Stomatitis (Gastrointestinal disorders) | 8 | 12
Vomiting (Gastrointestinal disorders) | 142 | 23
Asthenia (General disorders) | 44 | 12
Fatigue (General disorders) | 71 | 44
Influenza like illness (General disorders) | 12 | 7
Oedema peripheral (General disorders) | 22 | 24
Pyrexia (General disorders) | 37 | 43
Bronchitis (Infections and infestations) | 14 | 9
Influenza (Infections and infestations) | 17 | 7
Nasopharyngitis (Infections and infestations) | 20 | 16
Oral herpes (Infections and infestations) | 13 | 6
Rhinitis (Infections and infestations) | 13 | 4
Upper respiratory tract infection (Infections and infestations) | 32 | 32
Urinary tract infection (Infections and infestations) | 18 | 13
Fall (Injury, poisoning and procedural complications) | 14 | 4
Alanine aminotransferase increased (Investigations) | 12 | 4
Decreased appetite (Metabolism and nutrition disorders) | 31 | 15
Hypokalaemia (Metabolism and nutrition disorders) | 21 | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 45 | 32
Back pain (Musculoskeletal and connective tissue disorders) | 27 | 24
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28 | 12
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 115 | 126
Dizziness (Nervous system disorders) | 25 | 21
Headache (Nervous system disorders) | 25 | 26
Anxiety (Psychiatric disorders) | 17 | 8
Insomnia (Psychiatric disorders) | 22 | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 30 | 39
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 | 17
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 | 19
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 18
Hypertension (Vascular disorders) | 19 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/35/NCT01757535/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/35/NCT01757535/SAP_001.pdf